CLINICAL TRIAL: NCT00011492
Title: Evaluation for NIDCD Head & Neck Surgery Branch Clinical Research Protocols
Brief Title: Patient Evaluation for Head and Neck Surgery Branch Studies
Status: Terminated | Type: Observational
Why Stopped: Closed by Sponsor/Data Safety monitoring Board/IRB
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010099; 01-DC-0099; NCT00045071 (obsolete NCT alias)
Record Dates: First submitted 2001-02-22; First posted 2001-02-23 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-08

CONDITIONS: Head and Neck Neoplasms; Pharyngeal Cancer; Oral Cancer; Carcinoma, Squamous Cell; Laryngeal Cancer
Keywords: Oral Cancer; Squamous Cell Cancer; Head and Neck Cancer; Laryngeal Cancer; Pharnygeal Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Pharyngeal Neoplasms; Mouth Neoplasms; Carcinoma, Squamous Cell; Laryngeal Neoplasms; Neoplasms, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1/All Patients: All eligible patients

SUMMARY:
This purpose of this protocol is to evaluate and identify patients who may be eligible for actively enrolling NIH clinical research protocols for head and neck cancer; or provide standard evaluations and treatment necessary for patients with head and neck cancers enrolled in other NIH clinical protocols that do not include such treatment. Participants screened under this protocol will not be required to join a research study; the decision will be voluntary.

Patients with head and neck cancer may enroll in this study. Participants may undergo various tests, described below, to determine their eligibility for participation in a specific clinical trial. Other tests may also be required, depending on the protocol or treatment for which the patient is being considered:

* Blood tests About 3 to 5 tablespoons of blood will be drawn for routine tests, HLA typing and hepatitis and HIV screening.
* Magnetic resonance imaging (MRI) This imaging procedure uses a powerful magnetic field to produce pictures of parts of the body in small section views. The test does not use radiation and may be done with or without a contrast dye material.
* Computerized tomography (CT) This procedure uses x-rays to produces three-dimensional images of body organs in small section views. A contrast dye may or may not be used.
* Positron emission tomography (PET) PET scans allow the doctor to see the activity of cells in specific body tissues. It requires injection of a radioactive material that attaches to a sugar fluid. The fluid goes to very active cells, such as cancer cells, revealing tumors.
* Pulmonary function tests These tests use a machine the patient breathes into to measure the volume of air the patient can move in and out of the lungs.
* Arteriogram, or angiogram The anatomy of the blood vessels can be seen using this procedure, which involves placing a small catheter (plastic tube) into an artery and injecting a contrast solution. Special X-rays are then taken to show the blood vessels.
* Endoscopy This procedure is done to evaluate the mouth and throat. A tube with a light on the end and special fibers is inserted down the throat to allow the surgeon to examine the throat and, if needed, biopsy a piece of tissue for microscopic study. The test is usually done under general anesthesia in the operating room.
* Biopsy A piece of tissue or tumor is removed for examination under the microscope. When a biopsy is done in the neck area, a small amount of anesthetic is injected into the area of the biopsy. The biopsy may be done with 1) a small needle to pull out some tissue, 2) a cookie-cutter-like instrument to punch out a small piece of tissue, or 3) a small knife to cut out a piece of tissue. A knife biopsy may be done in the operating room or the clinic depending on the location of the biopsy and precautions required.

When the tests are done, the physician will discuss the results with the patient. Patients eligible for a research study will be offered participation. For those not eligible for a study, other therapies will be discussed and the patient will return to the care of his or her primary physician. In special circumstances, patients may be offered standard non-experimental treatment at NIH.

DETAILED DESCRIPTION:
This protocol will provide a means for screening potential candidates for NIDCD Head and Neck Surgery Branch (HNSB), and inter-institute protocols with NCI and NIDCR. No investigational treatments will be administered on this protocol. The Principal Investigator may, however, approve a patient who has been determined to be ineligible for investigational protocols to undergo standard treatment because they present a unique clinical experience for maintaining clinical skills of HNSB physicians and training of clinical fellows.

Background:

Potential research candidates are referred to the NIDCD HNSB by physicians and by patients themselves. Up to half of all research subjects now admitted to NIH protocols are self-referred. Each patient undergoes thorough telephone screening including a request for the results of outside laboratory tests, scans, x-rays and protocols. Some protocols may require additional diagnostic tests or that tests be repeated to obtain more current results in an effort to establish eligibility according to protocol specifications. The purpose of this protocol is to provide a means for patients to undergo: (1) evaluation to meet the eligibility requirements of active NIDCD HNSB and inter-institute protocols; and (2) standard treatment to ensure adequate expertise and training of surgeons and clinical associates and to provide an environment that stimulates ideas for clinical research.

Objectives:

-To permit evaluation of patients referred to the NIDCD Head and Neck Surgery Branch

(HNSB) in order to identify individuals who will be suitable candidates for HNSB

clinical research protocols and inter-institute protocols with NCI and NIDCR.

-To permit standard treatment in specific circumstances for patients not eligible for a

current investigational protocol, but who present a unique clinical training opportunity or

who present a clinical condition during screening that requires immediate intervention to

prevent compromise to the patient s well-being.

Eligibility:

Inclusion Criteria:

* Age 18 and older
* Patients at risk, suspected of having, or with a biopsy proven neoplastic disease of the

head and neck.

-Patient is able to provide informed consent.

Exclusion Criteria:

* Women who are pregnant are not eligible
* Candidates who do not meet the inclusion criteria.

Design:

-Patients enrolled on this protocol will be evaluated by NIDCD HNSB physicians to

determine the individual s suitability for participation in a clinical research protocol.

Specific clinical pathology and research diagnostic tests may be required to meet the

eligibility criteria of a protocol. These may include, but are not limited to:

* Blood tests
* Computerized Tomography scans without or with contrast
* Magnetic Resonance Imaging without or with gadolinium contrast
* Positron Emission Tomography
* Arterio- or Angiogram
* Nuclear Medicine scans (e.g. Technecium, Gallium)
* Pulmonary Function Tests
* Endoscopy of upper aerodigestive tract
* Fine needle aspiration or Tissue Biopsy

Other tests that are clinically indicated may be performed.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 18 and older

Patients at risk. Suspected of having, or with a biopsy proven neoplastic disease of the head and neck.

Patient is able to provide informed consent.

EXCLUSION CRITERIA:

Women who are pregnant and not eligible.

Candidates who do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Head and Neck Disorders including Cancer will be screened under this protocol. Subjects can be from any location, age 4 - no maximum age, any gender, race, and ethnicity. Subjects can selfrefer or come from another protocol or physician's office.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2001-03-12 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
To permit evaluation of patients to NIDCD Head and Neck Branch in order to identify suitable candidates for NIDCD NCI Head and Neck protocols or other NCI-based Head and Neck Cancer protocols. | 12/31/2021
  To evaluate patients to meet the eligibility criteria of active NIDCD HNSB or other IC Head and Neck protocols

SECONDARY OUTCOMES:
Evaluation of standard care treatment for subjects with head and neck disorders, train ENT surgeons and clinical associates in surgical intervention procedures and stimulate new ideas for clinical research | 12/31/2021
  To provide expertise clinical care during screening and surgical procedures and training of ENT and other Physicians and Clinical Associates in the care and surgical procedures needed for head and neck subjects and the development of new head and neck surgery and treatment protocols and procedures, along with new ideas for clinical HN research

CONTACTS AND LOCATIONS:
Overall Officials: Carter Van Waes, M.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2001-DC-0099.html